CLINICAL TRIAL: NCT05901948
Title: Asherman Syndrome: Pre-surgical Grading to Improve Gauge Prognostic Values and Improve Outcomes
Brief Title: Pre-Surgical Grading System of Asherman Syndrome
Status: Completed | Type: Observational
Sponsor: Ebtesama Hospital (Other)
Responsible Party: Principal Investigator, Yehia Shawki, Endoscopy unit director, Ebtesama Hospital
Other Study IDs: 100032023002
Record Dates: First submitted 2023-06-04; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Asherman Syndrome
Keywords: Asherman Syndrome; Hysteroscopy; Intra-Uterine Surgery; Intra-Uterine Adhesions; Classification
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asherman Patients: Patients diagnosed with Asherman syndrome based on patient complaint of hypomenorrhea or amenorrhea and hysterosalpingography.
  Interventions: Other: Classification

INTERVENTIONS:
Other: Classification — Novel Asherman Scoring Classification

SUMMARY:
Utilising a novel pre-surgical grading system to class cases of asherman syndrome into 3 groups based on expected difficulty of surgery and potential prognostic outcomes.

DETAILED DESCRIPTION:
Using the grading system, patients are classified into Mild, Moderate and Severe Asherman Syndrome. With the mild disease having the best prognostic value and a 1 step procedure, Moderate cases having a mediocre prognosis and usually multi-step procedure and Severe cases having a poor prognosis and counseled to other options. This observational study looks at the surgical outcomes following hysteroscopy for cases graded according to the new system to identify the accuracy of the classification in predicting the surgical success and prognostic value.

ELIGIBILITY:
Inclusion Criteria:

* Asherman Syndrome
* intra-uterine synechiae

Exclusion Criteria:

* patients with a fundectomy or uterine reduction surgery.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients complaining of hypomenorrhea, amenorrhea or infertility, who have a hysterosalpingography confirming intrauterine adhesions (Asherman Syndrome)
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Percentage Resumption of normal cavity on hystero-salpingography | 1 month
  assessing the improvement of the cavity of the uterus in hystero-salpingography

SECONDARY OUTCOMES:
Menses | 3 months
  Improvement in patients menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Osama Shawki, MD, Study Chair — Cairo University
Locations (1):
- Ebtesama Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Sharing IPD in an effort to garner more research and interest in the field
Supporting Information: Study Protocol
Time Frame: 1 year after completion

REFERENCES:
- [Result] Dreisler E, Kjer JJ. Asherman's syndrome: current perspectives on diagnosis and management. Int J Womens Health. 2019 Mar 20;11:191-198. doi: 10.2147/IJWH.S165474. eCollection 2019. PMID 30936754
- [Result] Salazar CA, Isaacson K, Morris S. A comprehensive review of Asherman's syndrome: causes, symptoms and treatment options. Curr Opin Obstet Gynecol. 2017 Aug;29(4):249-256. doi: 10.1097/GCO.0000000000000378. PMID 28582327
- [Result] Di Guardo F, Della Corte L, Vilos GA, Carugno J, Torok P, Giampaolino P, Manchanda R, Vitale SG. Evaluation and treatment of infertile women with Asherman syndrome: an updated review focusing on the role of hysteroscopy. Reprod Biomed Online. 2020 Jul;41(1):55-61. doi: 10.1016/j.rbmo.2020.03.021. Epub 2020 Apr 28. PMID 32444259